CLINICAL TRIAL: NCT07174726
Title: A Phase 2 Open-label Study to Evaluate the Safety of Laruparetigene Zovaparvovec Administered Bilaterally in Male Participants With X-Linked Retinitis Pigmentosa
Acronym: Landscape
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RPGR-005 Landscape
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: X-Linked Retinitis Pigmentosa (XLRP)
Keywords: XLRP; retinal degeneration; RPGR; adeno-associated virus; AAV; gene therapy
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: To evaluate the long-term safety and tolerability of laruparetigene zovaparvovec administered bilaterally via subretinal injection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants undergo pars plana vitrectomy and receive a central subretinal administration both eyes (Experimental): On Day 1, participants will undergo a pars plana vitrectomy and receive a central subretinal administration of laruparetigene zovaparvovec in their first treated study eye.
  For the first six participants, participants will undergo a pars plana vitrectomy followed by a central subretinal administration of laruparetigene zovaparvovec in their second eye between 30 and 60 days after the first surgery.
  Once the first six study participants have been dosed in both eyes, the interval between dosing of the first and second eye may be reduced to a minimum of 7 days (and up to 14 days) for up to four of the remaining participants enrolled in the study, provided the following conditions are met:
  * No unexpected safety concerns were observed following dosing of the first eye.
  * An independent safety review by the Sponsor, Investigator, and DSMC Chair confirms that bilateral dosing may proceed.
  Interventions: Biological: Adeno-associated virus vector expressing a human RPGR gene

INTERVENTIONS:
Biological: Adeno-associated virus vector expressing a human RPGR gene — Male participants 12-50 years of age treated by subretinal injection with the dose of AGTC-501

SUMMARY:
The purpose of this Phase 2 Study is to see if the investigational study drug, laruparetigene zovaparvovec, also known as AGTC-501, given in both eyes, is safe and works to preserve and/or improve vision and other symptoms of XLRP.

DETAILED DESCRIPTION:
XLRP is a genetic (inherited) eye disease that affects cells in the retina (the lining of the back of the eye that detects light). It causes night blindness and gradual worsening of your vision.

The purpose of this Phase 2 Study is to see if the investigational study drug, laruparetigene zovaparvovec, also known as AGTC-501, given in both eyes, is safe and works to preserve and/or improve vision and other symptoms of XLRP.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

* Provide written informed consent or assent (per local regulation) prior to the conduct of any study-related procedures. Participants who provide assent must have a parent, guardian, or legal representative provide written informed consent.
* Be between 12 and 50 years of age (inclusive) at the time of providing informed consent and assent (as applicable)
* Be male (XY chromosome) and have at least 1 documented pathogenic or likely pathogenic variant in the RPGR gene, within exons 1-14 and/or ORF15, from an appropriately certified or accredited laboratory
* Have a clinical diagnosis of XLRP
* Be in good general health to withstand subretinal surgery and perioperative medications based on a complete physical examination and results from hematology, chemistry, and coagulation analyses performed at screening
* Be able and willing, as assessed by the Investigator, to follow study instructions, complete study assessments, comply with the protocol, and attend all study visits
* If the participant has a parent or caregiver, the parent or caregiver must be able to follow study instructions, comply with the protocol, and attend study visits with the participant, as required

Ocular inclusion criteria (both eyes)

* Have a BCVA ≤ 78 letters (approximately Snellen, 20/32) and ≥ 34 letters (approximately Snellen, 20/200) in each eye based on an ETDRS chart at each screening visit. The ETDRS letter score is the main visual acuity inclusion criterion for participants. Participants unable to read the ETDRS letters may use a tumbling "E" chart for the BCVA assessments
* Have an LLVA ≤ 64 letters (approximately Snellen, 20/50) in both eyes based on an ETDRS chart at each screening visit. Participants unable to read the ETDRS letters may use a tumbling "E" chart for the LLVA assessments
* Have an LLD of >10 letters
* Be able to perform all tests of visual and retinal function and structure in both eyes based on the participant's reliability and fixation, per the Investigator's discretion
* Have a detectable mean macular sensitivity by MAIA microperimetry at baseline between 1 and 12 dB in both eyes, as determined by the Investigator and confirmed by the central reading center (CRC), with a fixation loss ≤ 20% at each screening visit
* Have a detectable sub-foveal EZ line as assessed by SD-OCT in both eyes as confirmed by the CRC

Exclusion Criteria:

General Exclusion Criteria

* Have other known disease-causing mutations documented in the participant's medical history or identified through a retinal dystrophy gene panel that, in the opinion of the Investigator, would interfere with the potential therapeutic effect of the study drug or the quality of the assessments
* For participants with herpes simplex virus (HSV):

  1. Have a history of oral or genital herpes and be unable and/or unwilling to use a prophylactic antiviral medication.
  2. Have a history of ocular herpes.
  3. Have active oral or genital herpes or are currently receiving treatment for active HSV infection
* Have complicating systemic diseases (e.g., medical conditions causing immunosuppression, autoimmunity, active systemic infection) that would preclude the gene transfer or ocular surgery if not adequately managed or treated
* Have a known sensitivity or allergy to systemic corticosteroids or other immunosuppressive medications
* Have used anticoagulant agents that may alter coagulation (e.g., warfarin, heparin, apixaban, or high-dose docosahexaenoic acid [fish oil]) within 7 days prior to study drug administration (ibuprofen, aspirin, or similar agents are acceptable
* Have received any vaccination/immunization within 60 days prior to Day 1 and/or during screening with the exception of the influenza vaccine, which is only exclusionary if received within 28 days prior to Day 1
* Have used systemic corticosteroids or other immunosuppressive medications within 3 months prior to study drug administration. Corticosteroids used on an as-needed basis administered by insufflation, inhalation, or local administration to the skin and mucosa such as Symbicort® (budesonide/formoterol), Flonase® (fluticasone propionate), and skin creams and ointments containing corticosteroids shall not be exclusionary
* If sexually active or planning to become sexually active, are unwilling to use barrier contraception for 3 months following study drug administration
* Have any other condition or reason that, in the opinion of the Investigator, would prevent the participant from completing all study assessments
* Have any other condition or reason that, in the opinion of the Investigator, makes the participant unsuitable for the study
* Are currently participating or recently participated in any other research protocol involving investigational agents or therapies that, in the opinion of the Investigator, would make the participant unsuitable for the study. Recent participation is defined as participation within 90 days of initial screening for this study OR within 10 half-lives of the investigational drug, whichever is longer
* Have previously received any adeno-associated virus (AAV) gene therapy product, stem cell therapy, cell-based therapy, or similar biologics

Ocular exclusion criteria (either eye)

* Have pre-existing eye conditions in either eye that would preclude the planned surgery, interfere with the interpretation of study endpoints, or increase the risk of surgical complications (e.g., corneal opacities, diabetic retinopathy, retinal vasculitis, glaucoma, active cystoid macular edema)
* Have significant media opacity impacting evaluation of the retina or vitreous in either eye. This includes cataracts considered to be a major contributor to reducing visual acuity and/or if the participant is likely to require cataract extraction within 3 months of study drug administration
* Had intraocular surgery in either eye within the 90 days prior to the planned administration of study drug
* Have any active ocular/intraocular infection or inflammation (e.g., severe blepharitis, infectious conjunctivitis, keratitis, scleritis, endophthalmitis, idiopathic or autoimmune-associated uveitis, or herpetic lesions) in either eye
* Have a history of corticosteroid-induced raised intraocular pressure (IOP) of > 25 mmHg following corticosteroid exposure in either eye, despite topical IOP-lowering pharmacologic therapy
* Have any artificial retinal implant or prosthesis in either eye
* Have an absence of clear ocular media and/or inadequate pupil dilation to facilitate good quality SD-OCT images in either eye.
* Have any history of rhegmatogenous retinal detachment in either eye
* Have myopia (spherical equivalent) exceeding -10 diopters Investigator or the presence of pathologic myopia in either eye.

Ages: 12 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 10 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-12-15 (Estimated)

PRIMARY OUTCOMES:
The number and percentage of participants experiencing Grade 3 or higher ocular or non-ocular treatment-emergent adverse events (TEAEs), including treatment-emergent serious adverse events (SAEs), at Month 12 | Day 0 - Month 12

SECONDARY OUTCOMES:
The number and percentage of participants experiencing ocular or non-ocular TEAEs, including treatment-emergent SAEs during the Study period | Day 0-5 years
Change from baseline in low-luminance visual acuity (LLVA) using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity at Month 12 | Day 0 - Month 12
Change from baseline in mean sensitivity across the whole grid, as measured by macular integrity assessment (MAIA) microperimetry at Month 12 | Day 0 - Month 12
Response, as measured by MAIA microperimetry, where response is defined as a ≥ 7 dB visual sensitivity improvement from baseline in at least 5 loci at Month 12 | Day 0 - Month 12
Change from baseline in full-field stimulus threshold (FST) at Month 12 | Day 0 - Month 12
Change from baseline in best-corrected visual acuity (BCVA) using ETDRS visual acuity at Month 12 | Day 0 - Month 12
Change from baseline in low-luminance deficit using ETDRS visual acuity at Month 12 | Day 0 - Month 12
Proportion of responding eyes at Month 12 where responder is defined as an improvement of at least 15 letters on LLVA | Day 0 - Month 12
Change from baseline in ellipsoid zone (EZ) area measured by spectral domain-optical coherence tomography (SD-OCT) at Month 12 | Day 0 - Month 12
Change from baseline in 7 domain scores from a Michigan Retinal Degeneration Questionnaire (MRDQ) at Month 12 | Day 0 - Month 12
Change from baseline in the Mobility Standardized Test-Virtual Reality (MOST-VR) course test score at Month 12 | Day 0- Month 12

CONTACTS AND LOCATIONS:
Overall Officials: None None, Principal Investigator
Locations (6):
- United States (6):
  - University of Florida Jacksonville Ophthalmology, Jacksonville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Duke Eye Center, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - OHSU Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No